CLINICAL TRIAL: NCT06412575
Title: Joint Nasogastric Tube (JNT) Versus Traditional Decompression Nasogastric Tube (TNT) to Guided OGT-overlap Oesophagojejunostomy in Laparoscopic Total Gastrectomy: A Randomized Controlled Trial
Brief Title: JNT Versus TNT to Guided OGT-overlap Oesophagojejunostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2024-142
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Gastric/Gastroesophageal Junction (g/Gej) Cancer
Keywords: Gastric tumor; Gastric/gastroesophageal junction (G/GEJ); Laparoscopic total gastrectomy; Overlap anastomosis; Joint nasogastric tube
MeSH Terms: conditions — Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: This study was a parallel, open-label randomized trial that aimed to assess safety and efficiency of JNT and TNT to guided OGT-overlap oesophagojejunostomy. Gastric/gastroesophageal junction (G/GEJ) cancer patients who underwent LTG with OGT-overlap oesophagojejunostomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JNT group (Experimental): In the JNT group, the Joint Nasogastric Tube (JNT) was put into the oesophageallumen from the nose, to guide the cutting of a small enterotomy on the posterior oesophageal stump.
  Interventions: Procedure: JNT Guided OGT-overlap Oesophagojejunostomy
- TNT group (Active Comparator): In the TNT group, the traditional decompression nasogastric tube (TNT) was put into the oesophageallumen from the nose, to guide the cutting of a small enterotomy on the posterior oesophageal stump.
  Interventions: Procedure: TNT Guided OGT-overlap Oesophagojejunostomy

INTERVENTIONS:
Procedure: JNT Guided OGT-overlap Oesophagojejunostomy — In the JNT group, the Joint Nasogastric Tube (JNT) was put into the oesophageallumen from the nose, to guide the cutting of a small enterotomy on the posterior oesophageal stump.
  Arms: JNT group
Procedure: TNT Guided OGT-overlap Oesophagojejunostomy — In the TNT group, the Traditional Decompression Nasogastric Tube (TNT) was put into the oesophageallumen from the nose, to guide the cutting of a small enterotomy on the posterior oesophageal stump.
  Arms: TNT group

SUMMARY:
Gastric/gastroesophageal junction (G/GEJ) cancer patients who underwent laparoscopic total gastrectomy (LTG) were eligible for this study

DETAILED DESCRIPTION:
All patients enrolled in our study underwent standard laparoscopic total gastrectomy (LTG) with D2 lymphadenectomy and OGT-overlap oesophagojejunostomy according to the Japanese Gastric Cancer Association treatment guidelines and our previous reports. When the surgeons decided to perform OGT-overlap oesophagojejunostomy after gastrectomy, we randomised the patients into the Traditional Decompression Nasogastric Tube (TNT) group or Joint Nasogastric Tube (JNT) group by simple randomization operatively.

In the TNT group, the TNT was put into the oesophageallumen from the nose, to guide the cutting of a small enterotomy on the posterior oesophagealstump . While in the JNT group, the JNT was used to substitute the TNT. After the anastomosis was completed, the team of surgeons performed an intraoperative gastroscopy to check for defects, bleeding, and stenosis in the anastomosis, and esophageal pseudocanals, and also to confirm whether the esophageal mucosa was damaged by TNT or JNT.

ELIGIBILITY:
Inclusion Criteria:

(1) Age 18-75 years; (2) Physical status score (ECOG) 0-2 points; (3) Preoperative pathological examination to diagnose gastric/gastroesophageal junction (G/GEJ) cancer; (4)No obvious contraindications for surgery; (5)Did not found metastasis preoperatively and intraoperatively; (6)Confirmed tumours invade oesophagus no more than 3cm intraoperatively; (7) Expected to perform OGT-overlap oesophagojejunostomy after lymphadenectomy and gastrectomy in the operation of laparoscopic total gastrectomy.

Exclusion Criteria:

(1)Underwent radiotherapy for G/GEJ cancer preoperatively; (2) continuous HIPEC after operation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Time of OGT and nasogastric tube (NT) connection | Surgery
  Time starts from insertion of the NT through the nose, to the end of the NT docking with the OGT and successfully implanted into the esophageal cavity.

SECONDARY OUTCOMES:
Time of nasogastric tube (NT) insertion | Surgery
  Time starts from insertion of the NT through the nose, to the front end of the NT reaching the esophageal stump.
Time of oesophagojejunostomy | Surgery
  Time starts from making the entry hole for the anastomosis on the oesophagealstump, to the end of the common entry hole was closed using barbed threads.

OTHER OUTCOMES:
Oesophageal mucosal injury | Surgery
  the oesophagealmucosa is observed endoscopically after the common hole is closed. Patients with esophageal mucosal injury can be shown as esophageal mucosal surface with mucosal injury caused by nasogastric tube (NT) .
)Inserting anvil fork into oesophageallumen at first attempt | Surgery
  when inserting the anvil fork into the oesophagealhole, the anvil fork can be correctly placed in a satisfactory position and at a satisfactory angle into the oesophagealmucosa canal to be fired for oesophagojejunostomy by inserting it only once.
Inserting NT to oesophagealstump at first attempt | Surgery
  when inserting the NT from nose to the oesophagealstump only once without pulling out and reinserting.
Early postoperative complications | Within 30 days after the surgery
  postoperative complications were assessed within 30 days after the surgery and rated following Clavien-Dindo classification (CDC) system

CONTACTS AND LOCATIONS:
Overall Officials: Xinhua Chen, Ph.D, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
If other researchers are interest in the IPD, please contact Xinhua Chen(xinhuachen03@163.com）.